CLINICAL TRIAL: NCT04352153
Title: A Randomized, Prospective, Controlled Study of the Efficacy and Safety of Uralyt-U Combined With Febuxostat in the Treatment of Hyperuricemia With Uric Acid Stones
Brief Title: Role of Uralyt-U in Patients With Hyperuricemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ai Peng (Other)
Responsible Party: Sponsor-Investigator, Ai Peng, Director of the department of Nephrology, Shanghai 10th people's hospital, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uralyt-U
Record Dates: First submitted 2020-04-10; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Uric Acid Stones; Hyperuricemia
Keywords: Uric Acid Stones; Hyperuricemia; Uralyt-U
MeSH Terms: conditions — Hyperuricemia | interventions — Febuxostat; Citrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-use group (Experimental): Febuxostat is taken at a dose of 20 mg once a day. During the medication period, the urine pH of each subject is monitored and recorded in the morning, noon and night.
  Interventions: Drug: Febuxostat
- Research group (Experimental): Febuxostat is taken at a dose of 20 mg once a day, potassium sodium hydrogen citrate granules 7.5 g / day, 2.5 g / per time, three times a day. During the medication period, the urine pH of each subject is monitored and recorded in the morning, noon and night.
  Interventions: Drug: Febuxostat; Drug: Uralyt-U

INTERVENTIONS:
Drug: Febuxostat — Febuxostat is taken at a dose of 20 mg once a day. During the medication period, the urine pH of each subject is monitored and recorded in the morning, noon and night.
  Other Names: Uloric; Adenuric
Drug: Uralyt-U — Febuxostat is taken at a dose of 20 mg once a day, potassium sodium hydrogen citrate granules 7.5 g / day, 2.5 g / per time, three times a day. During the medication period, the urine pH of each subject is monitored and recorded in the morning, noon and night.
  Other Names: potassium sodium hydrogen citrate granules
  Arms: Research group

SUMMARY:
The purpose of the study is to provide a more direct and objective basis for the widespread use of potassium sodium hydrogen citrate granules in the treatment of uric acid stones.

DETAILED DESCRIPTION:
Hyperuricemia (HUA) is a common systemic metabolic disease. Its incidence is increasing year by year and more young people suffer from hyperuricemia. HUA can not only cause the onset of gouty arthritis, and then affect joint function, and even cause joint deformities. It can also cause damage to multiple organs such as the heart, brain, and kidney through multiple channels. Chronic kidney disease (CKD) refers to chronic kidney structural and dysfunction caused by various reasons. HUA is an independent risk factor that accelerates the progress of CKD. Studies have shown that lowering uric acid is another key treatment to delay the progress of CKD. A large number of studies have shown that the formation of uric acid crystals is the main mechanism of inducing renal injury.

In 2017, the "Multidisciplinary Expert Consensus for the Diagnosis and Treatment of Hyperuricemia-Related Diseases in China" recommended that patients with hyperuricemia receiving uric acid lowering drugs, especially those treated with uric acid excretion drugs and patients with uric acid nephrolithiasis, recommended that the pH of urine be adjusted during pH6.2 ~ 6.9 to increase the solubility of uric acid in urine. It is recommended to use sodium bicarbonate or potassium sodium citrate drugs to alkalinize urine, but it is not clear if there is any difference in the kinetic parameters of urine alkalinity, compliance rate of alkalinized urine and safety between sodium bicarbonate and potassium sodium citrate. No "head-to-head" clinical publications have been reported. This clinical trial was designed to evaluate the rate of alkalinization of urine, the therapeutic effect of renal lithiasis and adverse reactions between the sodium bicarbonate and potassium sodium hydrogen citrate granules in healthy people and patients with hyperuricemia and renal calculi (uric acid). This study provides a more direct and objective basis for the widespread use of potassium sodium hydrogen citrate granules in the treatment of uric acid stones.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old, male, outpatient or inpatient;
* Acidic urinary stones
* Serum uric acid value ≥480 µmol / L;
* Other concomitant diseases (such as hypertension, hyperlipidemia, diabetes, etc.) are in a stable condition, and the dosage of other diseases is not changed during the test.
* eGFR≥30ml / min;

Exclusion Criteria:

* Pregnant or lactating women;
* Patients with acute or chronic renal failure (eGFR <30ml / min);
* Patients with severe liver dysfunction (ALT, AST≥70 IU);
* In patients with uncontrolled hypertension, systolic blood pressure ≥160 and / or diastolic blood pressure ≥110mmHg;
* In uncontrolled diabetic patients, fasting blood glucose is> 10mmol / L, and / or glycated hemoglobin is ≥9%;
* Patients that are taking atorvastatin, losartan, amlodipine, fenofibrate, pyrazinamide, tincture diuretics, thiazide diuretics, glucocorticoids, immunosuppressive agents and other drugs that affect uric acid excretion Drugs, those taking aspirin at a dose of> 325mg / day;
* Cancer patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Uric acid stones | 3 months
  Uric acid stones will be estimated by dual-source CT examination
Uric acid stones | 6 months
  Uric acid stones will be estimated by dual-source CT examination

SECONDARY OUTCOMES:
Blood uric acid | 1 month
  Blood uric acid will be detected
Blood uric acid | 3 months
  Blood uric acid will be detected
Blood uric acid | 6 months
  Blood uric acid will be detected

CONTACTS AND LOCATIONS:
Overall Officials: Ai Peng, Ph.D., M.D., Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Department of Nephrolgoy, Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xue W, Cheng J, Zhao J, Wang L, Peng A, Liu X. Comparison potassium sodium hydrogen citrate with sodium bicarbonate in urine alkalization: a prospective crossover-controlled trial. Int Urol Nephrol. 2023 Jan;55(1):61-68. doi: 10.1007/s11255-022-03387-y. Epub 2022 Oct 19. PMID 36261757